CLINICAL TRIAL: NCT00686101
Title: Knowledge and Perception of Smoking Risks/Consequences, Smoking Habits and Motivators for Smoking Cessation Among People With Schizophrenia
Brief Title: Knowledge and Perception of Smoking Risks/Consequences
Acronym: SmokCess
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Deanna Kelly, Deanna L. Kelly, Pharm.D., BCPP, Cheif Treatment Research Program, University of Maryland, Baltimore
Other Study IDs: HP-00042643; NIDA #425
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Cigarette Smoking; Schizophrenia
Keywords: Perception of risk; Smoking risks; Smoking consequences; Quitting smoking; Motivation to quit smoking; Schizophrenia
MeSH Terms: conditions — Cigarette Smoking; Schizophrenia; Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Normal control subjects (Males and females between 18-65 years, who smoke cigarettes daily, have an expired CO measurement of > 8 ppm to confirm cigarette smoking, who are not actively trying to quit smoking at the time of the interview, and who must be free from Axis I psychotic disorder.)
- 2: Subjects with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder (Males and females between 18-65 years, who smoke cigarettes daily, have an expired CO measurement of > 8 ppm to confirm cigarette smoking, and who are not actively trying to quit smoking at the time of the interview.)

SUMMARY:
This proposed 2-year questionnaire study examines views and attitudes regarding health risks of cigarette smoking, smoking patterns and motivators for cessation in smokers who suffer from schizophrenia compared to a sample of smokers without a major psychotic disorder.

DETAILED DESCRIPTION:
This proposed 2-year questionnaire study examines views and attitudes regarding health risks of cigarette smoking, smoking patterns and motivators for cessation in smokers who suffer from schizophrenia compared to a sample of smokers without a major psychotic disorder. The specific goals of this study are to 1) examine differences in the perceived consequences of smoking, smoking habits, and motivation to quit between adults with and without schizophrenia and 2) identify clinical and demographic variables (e.g., age, race, sex, age of smoking onset, knowledge of smoking consequences, insurance status, family support, co-occurring substance abuse, education level, current health status) associated with motivation to quit smoking among individuals with and without schizophrenia. This secondary goal is exploratory in nature. We will identify potential predictors in each group separately and also assess if these potential predictors differ between groups.

The study will consist of one 2-hour visit, where each subject, after signing consent, will participate in a semi-structured interview as well as answer clinical and demographic information. Patient volunteers will be recruited from the MPRC Outpatient and Inpatient Programs and through NIDA. Control subjects will be recruited by MPRC and NIDA via newspaper advertisements from the Baltimore metropolitan area. We anticipate recruiting up to 110 schizophrenia patients for a total of 100 completers and up to 110 normal controls for a total of 100 completers. All participants will be 18-65 years old, will smoke cigarettes daily, and must not be interested in reducing or quitting tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18-65 years
* Minimum of 5 cigarettes daily.
* Expired CO measurement of > 8 ppm to confirm cigarette smoking
* For the schizophrenia group, must have a DSM-IV diagnosis of schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* For the normal control group, must be free from Axis I psychotic disorder. (other psychiatric comorbidity will not be excluded)
* For all subjects, anyone actively trying to quit smoking at the time of the interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient volunteers will be recruited from the MPRC Outpatient and Inpatient Programs and through NIDA. Control subjects will be recruited by MPRC and NIDA via newspaper advertisements from the Baltimore metropolitan area. We anticipate recruiting up to 110 schizophrenia patients for a total of 100 completers and up to 110 normal controls for a total of 100 completers. All participants will be 18-65 years old, will smoke cigarettes daily, and must not be interested in reducing or quitting tobacco use. Nicotine dependence appears to be about equally represented among ethnic and racial backgrounds and gender.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The measure will be the differences in smoking perceptions/risk and motivation as assessed by the questionnaires between smokers with and without schizophrenia. | For each subject, the time frame primarily evaluated will be the length of his or her use of cigarettes, primarily (but the time frame may be extended to include other evaluated factors, such as education or family/economic support).

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, PharmD, BCPP, Principal Investigator — University of Maryland, College Park; Steve Heishman, MD, Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - National Institute on Drug Abuse (Johns Hopkins Bayview Campus), Baltimore, Maryland
  - Maryland Psychiatric Research Center, University of Maryland School of Medicine, Baltimore, Maryland